CLINICAL TRIAL: NCT06676410
Title: Clinical Trial to Evaluate the Efficacy and Safety of Codivir® in Addition to Standard Antiretroviral Treatment for HIV Infection in Antiretroviral-naïve Participants
Acronym: Codivir®
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Code Pharma (Industry)
Collaborators: Galilee CBR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-22-03
Record Dates: First submitted 2024-10-01; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: HIV; HIV Infection
Keywords: HIV; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Demography; Body Height; Body Mass Index; Pregnancy Tests; Random Allocation; Anti-Retroviral Agents

STUDY DESIGN:
Intervention Model Description: Randomization
  Forty participants with a recent diagnosis of HIV infection, without previous antiretroviral treatment and indication to start antiretroviral treatment, will be randomized as follows:
  * 20 participants will receive Standard Antiretroviral Treatment + Codivir
  * 20 participants will only receive Standard Antiretroviral Treatment A randomization will be balanced by sex and age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Codivir® (Experimental): The study will begin with a two-week lead-in period (W-2 and W-1), when participants randomized to Codivir® will receive Codivir® 2 mL, 1 subcutaneous injection every day. Participants randomized to Standard Antiretroviral Treatment will wait for the next step.
  In Weeks 0-24, all participants will receive:
  * Single solid formulation (in 1 tablet) 1x/day with:
    * Tenofovir (TDF) 300 mg
    * Lamivudine (3TC) 300 mg
  * Darunavir (DRV) 800 mg, 1x/day
  * Ritonavir (RTV) 100 mg, 1x/day From V0 (W0, D0) to V6 (W12, D84) participants randomized to Codivir® will receive Codivir® as complementary therapy to the above antiretrovirals on alternate days (every other day).
  At V6 (week 12) treatment with Codivir® will end.
  Interventions: Other: ICF; Behavioral: Eligibility Assessment; Other: Demographic data; Diagnostic Test: Weight, height and BMI; Other: Vital Signs; Diagnostic Test: Medical evaluation; Diagnostic Test: Safety exam; Diagnostic Test: Pregnancy test; Diagnostic Test: Serology; Other: Randomization; Diagnostic Test: Apoptosis markers; Diagnostic Test: Cell activation markers; Diagnostic Test: Inflammation markers; Diagnostic Test: Proviral DNA:; Diagnostic Test: HIV-specific antibodies; Diagnostic Test: HIV viral load (RNA); Behavioral: Codivir® Training; Drug: Dispensing Codivir®; Other: Codivir® Accounting; Other: Concomitant medication; Other: Adverse events
- Antiretrovirals (ARTs) (Active Comparator): In Weeks 0-24, all participants will receive:
  * Single solid formulation (in 1 tablet) 1x/day with:
    * Tenofovir (TDF) 300 mg
    * Lamivudine (3TC) 300 mg
  * Darunavir (DRV) 800 mg, 1x/day
  * Ritonavir (RTV) 100 mg, 1x/day
  Interventions: Other: ICF; Behavioral: Eligibility Assessment; Other: Demographic data; Diagnostic Test: Weight, height and BMI; Other: Vital Signs; Diagnostic Test: Medical evaluation; Diagnostic Test: Safety exam; Diagnostic Test: Pregnancy test; Diagnostic Test: Serology; Other: Randomization; Diagnostic Test: Apoptosis markers; Diagnostic Test: Cell activation markers; Diagnostic Test: Inflammation markers; Diagnostic Test: Proviral DNA:; Diagnostic Test: HIV-specific antibodies; Diagnostic Test: HIV viral load (RNA); Other: Concomitant medication; Other: Adverse events; Drug: Antiretrovirals

INTERVENTIONS:
Other: ICF — Application of Informed Consent Form.
Behavioral: Eligibility Assessment — Assessment of inclusion, exclusion and discontinuation criteria.
Other: Demographic data — Collection of demographic data.
Diagnostic Test: Weight, height and BMI — Weight and height measurement and body mass index calculation.
Other: Vital Signs — HR, BP and FR and T°, in addition to oximetry.
Diagnostic Test: Medical evaluation — Medical history and physical examination at screening. In other consultations, the medical evaluation is focused on viral load, CD4+ and new complaints.
Diagnostic Test: Safety exam — Blood collection for safety laboratory exams. Blood count, Na, K, U, C, amylase, total cholesterol and fractions, triglycerides, coagulation tests (TTTP, TT, platelets), TGO, TGP, AP, GGT, glycated hemoglobin, total bilirubin and fractions, creatine kinase and CKmB and urine I.
Diagnostic Test: Pregnancy test — β-HCG in urine in non-sterile women
Diagnostic Test: Serology — HBV (HBsAg, Anti-HBc) and HCV (anti-HCV-Ab).
Other: Randomization — Assignment to the Standard Antiretroviral Treatment + Codivir® group or the Standard Antiretroviral Treatment only group
Diagnostic Test: Apoptosis markers — Caspases and Annexin V.
Diagnostic Test: Cell activation markers — PBMCs will be isolated by density gradient centrifugation. The cells will then be tested for CD4+, CD8+, CD38 and HLA DR
Diagnostic Test: Inflammation markers — ultrasensitive CRP, D-dimer.
Diagnostic Test: Proviral DNA: — Total HIV DNA will be measured to estimate the size of the viral reservoir throughout the preparation.
Diagnostic Test: HIV-specific antibodies — Anti-HIV-1 specific antibody titers in plasma.
Diagnostic Test: HIV viral load (RNA) — Performed on plasma.
Behavioral: Codivir® Training — The participant is trained to self-inject Codivir®
  Arms: Codivir®
Drug: Dispensing Codivir® — the participant receives Codivir®
  Arms: Codivir®
Other: Codivir® Accounting — The Codivir® used since the last visit is accounted for
  Arms: Codivir®
Other: Concomitant medication — Record of concomitant medications used.
Other: Adverse events — Collection and recording of adverse events.
Drug: Antiretrovirals — Tenofovir - inhibits HIV-1 reverse transcriptase activity by competing with the natural substrate, deoxyadenosine 5'-triphosphate and, upon incorporation into DNA, causes DNA chain termination.
  * Lamivudine - potent selective inhibitor of HIV-1 and HIV-2 replication in vitro.
  * Darunavir - prevents the formation of mature infective viral particles, indicated for the treatment of the human immunodeficiency virus (HIV), which causes AIDS.
  * Ritonavir: antiretroviral protease inhibitor, widely used in combination with other protease inhibitors in the therapy and prevention of HIV infection, which causes the syndrome acquired immunodeficiency (AIDS).
  * Single solid formulation (in 1 tablet) 1x/day with:
  * Tenofovir (TDF) 300 mg
  * Lamivudine (3TC) 300 mg
  * Darunavir (DRV) 800 mg, 1x/day
  * Ritonavir (RTV) 100 mg, 1x/day
  Arms: Antiretrovirals (ARTs)

SUMMARY:
The study will begin with a two-week lead-in period (W-2 and W-1), when participants randomized to Codivir® will receive Codivir® 2 mL, 1 subcutaneous injection every day. Participants randomized to Standard Antiretroviral Treatment will wait for the next step.

At V0 (W0, D0) all participants will start the antiretroviral treatment described above.

From V0 (W0, D0) to V6 (W12, D84) participants randomized to Codivir® will receive Codivir® as complementary therapy to the above antiretrovirals on alternate days (every other day).

At V6 (W12, D84) treatment with Codivir® will end. At V7 (W24, D168) participation in the study will end. Viral load will be monitored during the study. In case of failure, participation in the study will be discontinued and the participant will be referred to receive the best treatment available for their case.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex;
2. Age ≥ 18 years;
3. HIV infection confirmed by serology (Ab for HIV1/HIV2) and HIV1/HIV2 RNA test;
4. Naive for antiretroviral treatment;
5. Viral load > 1,000 and < 50,000 copies/mL;
6. CD4 T lymphocyte (CD4) cell count >350 cells/mm3;
7. Body weight at V -1 > 50 Kg;
8. Signature of the ICF.

Exclusion Criteria:

1. Pregnancy, lactation or plan to become pregnant;
2. BMI < 18.5 kg/m2 at screening;
3. Coinfection with HBV (HBSAg +) or HCV;
4. Any Grade 3 or 4 clinically significant abnormality according to the Division of AIDS (DAIDS)* rating scale;
5. Any significant acute illness within 1 week before V0.
6. Use of any immunomodulatory therapy (including interferon), systemic steroids, or systemic chemotherapy within 4 weeks of screening;
7. Active malignancy or ongoing malignancy;
8. Changes in safety tests: neutrophil count < 1000 u/L; Hb < 9.0 gm/dl; platelet < 75,000 u/L; creatinine > 1.5 mg/dl, direct bilirubin > 85 μmol/l, AST or ALT > 2.5 X ULN;
9. Potential allergy or hypersensitivity to components of the Codivir® formulation.
10. Participation in another clinical trial within 12 months of screening.
11. Any medical condition that makes the participant unsuitable for the study or increases the risk of participation at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Variation between V-2 (baseline) and V6 (W12) in relation to the following parameter: • Estimated viral reservoir size by total blood proviral DNA. | 12 weeks
Variation between V-2 (baseline) and V6 (W12) in relation to the following parameter: CD4+ blood count | 12 weeks

SECONDARY OUTCOMES:
Variation between baseline visit and visit 7 (W24) in relation to the following parameter : Estimated viral reservoir size by total proviral DNA | 24 weeks
Variation between baseline visit and visit 7 (W24) in relation to the following parameter : CD4+ count. | 24 weeks
Variation between baseline visit and visit 7 (W24) in relation to the following parameter: apoptosis markers | 24 weeks
Variation between baseline visit and visit 7 (W24) in relation to the following parameter : Cell activation markers | 24 weeks
Variation between baseline visit and visit 7 (W24) in relation to the following parameter: Inflammation markers | 24 weeks
Variation between baseline visit and visit 7 (W24) in relation to the following parameter: Quantitative Proviral (DNA) | 24 weeks
Variation between baseline visit and visit 7 (W24) in relation to the following parameter: HIV viral load (RNA) | 24 weeks
- Comparison of viral load curves from all visits between the two groups. | 24 weeks
Codivir® safety by comparison of treatment-emergent adverse events in both groups. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- RDSS Research Center, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No